CLINICAL TRIAL: NCT05726786
Title: The Role of Preoperative Immunonutrition on Morbidity and Immune Response After Cystectomy - A Multicenter Randomized Controlled Trial (INCyst Trial)
Brief Title: The Role of Preoperative Immunonutrition on Morbidity and Immune Response After Cystectomy (INCyst Trial)
Acronym: INCyst
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Vaudois (Other)
Collaborators: Insel Gruppe AG, University Hospital Bern (Other); Hôpital Riviera-Chablais, Vaud-Valais (Other); University Hospital, Geneva (Other)
Responsible Party: Principal Investigator, Ilaria Lucca, MD, Principal Investigator, Centre Hospitalier Universitaire Vaudois
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: INCyst
Record Dates: First submitted 2023-01-16; First posted 2023-02-14 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Bladder Cancer; Interstitial Cystitis; Painful Bladder Syndrome; Neurogenic Bladder; Hemorrhagic Cystitis; Endometriosis; Bladder Disease
Keywords: Cystectomy; Immunonutrition; Complication; Malnutrition
MeSH Terms: conditions — Urinary Bladder Neoplasms; Cystitis, Interstitial; Urinary Bladder, Neurogenic; Cystitis, Hemorrhagic; Endometriosis; Urinary Bladder Diseases; Malnutrition | interventions — Immunonutrition Diet

STUDY DESIGN:
Intervention Model Description: Multicenter, prospective, controlled, pragmatic, parallel-group comparative study with block randomization stratified by centers
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Immunonutrition (Experimental): Seven days of preoperative oral supplementation with an immune-enhanced oral nutrition
  Interventions: Drug: Immunonutrition
- No immunonutrition (control) (No Intervention): Standard of care

INTERVENTIONS:
Drug: Immunonutrition — Immunonutrition: Oral Impact®, Nestlé Health Science, Switzerland.
  IN will be administered as per manufacturer suggestion, i.e. three times a day during 7 days preoperatively. Oral Impact® is a powdered oral feed that provides 309 kcal/bag
  Arms: Immunonutrition

SUMMARY:
The goal of this clinical trial research study is to evaluate the impact of preoperative oral immunonutrition (IN) on post-operative complications in patients undergoing a cystectomy.

As a secondary focus, this study will aim to develop a signature that would identify patients that would benefit the most from IN.

This is a multicentric (Swiss: N=3), prospective, controlled, pragmatic, parallel-group comparative study with block randomization stratified by centers.

DETAILED DESCRIPTION:
Despite standardized surgical technique and the development of new perioperative care protocols, cystectomy morbidity remains a serious challenge for urologists. Most common postoperative complications, such as infections, often lead to longer length of stay and worse survival. Malnutrition has been identified as an independent and modifiable risk factor for both mortality and morbidity. Immunonutrition (IN), containing arginine, ribonucleic acid and omega-3 polyunsaturated fatty acids, aims to improve the nutritional status, immunological function and clinical outcome of surgical patients. Meta-analyses have demonstrated that preoperative IN reduces complications and length of hospital stay after major bowel surgery. Evidence-based data on preoperative oral IN support for cystectomy patients are lacking, which does not allow this treatment to be widely accepted, recommended, or reimbursed by health insurances in most European countries. Uncertainties also remain about the exact mechanism by which IN modulates the host immune response.

Complication rates after cystectomy range from 40-75%. Malnutrition has been identified as an independent and modifiable risk factor for both mortality and morbidity. To date, and in the last 20 years, no single intervention has allowed for a significant reduction in morbidity after cystectomy, which remains one of the highest in surgery. The present adequately powered multicenter RCT has the potential of changing current practice by recommending preoperative IN before cystectomy in case of positive results. If the present RCT demonstrates a benefit in administrating IN prior to cystectomy, urological guidelines will be modified accordingly to this new evidence. IN will then be recommended before cystectomy for the patient's benefit. The investigators truly believe that the proposed study is of high clinical importance with potential impact on perioperative urology guidelines.

ELIGIBILITY:
Inclusion Criteria:

* Patient undergoing open cystectomy (for all reasons)
* Age ≥18 years
* Ability and willingness to provide informed consent documented by signature

Exclusion Criteria:

* Contraindications to IN, e.g. known hypersensitivity or allergy to lactose, fish oil or soy lecithin
* Severe diarrhoea requiring medical attention
* Current treatment with any immunosuppressive drug
* In standard practice, pregnant or lactating women are systematically rejected by the surgeon for this surgical procedure. Furthermore, during the pre-surgical anaesthesia consultation, the eligibility of each patient for anaesthesia will be assessed according to the usual criteria and recommendations of the anaesthesia service of the CHUV
* Other clinically significant concomitant disease affecting immunity (e.g., severe renal failure, HIV, SLE, transplant recipient, ...)
* Inability to follow the procedures of the study, e.g. due psychological disorders, dementia, etc.
* Participation in another study with investigational drug within the 30 days preceding and during the present study
* Previous enrolment into the current study
* Use of IN independently of the study
* Enrolment of the investigator, his/her family members, employees and other dependent persons
* Emergency procedure (less than 7 days between screening and surgery)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 232 (Estimated)
Dates: Start 2023-04-10 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Infectious complication after cystectomy | 30-days afetr surgery
  Determination of infectious complications rate at 30 days after surgery (pneumonia, urinary tract infection, surgical site infection, sepsis, shock).

SECONDARY OUTCOMES:
Comprehensive Complication Index (CCI) | 30 and 90 days after surgery
  Determination of the Comprehensive Complication Index (CCI) at 30 and 90 days after surgery. The range is between 0 (no complication) to 100 (death).
Mortality rate | 30 and 90 days after surgery
  Determination of the mortality rate at 30 and 90 days after surgery
Complication-free survival rate | 90-days after surgery
  Determination of the post-operative complication-free survival
Treatment compliance rate | Between Day -30 and Day -10 and at preoperative admission after intake of the allocated nutrition (Day -1)
  Serum arginine levels will be assessed at enrolment (between Day -30 and Day -10) and at preoperative admission after intake of the allocated nutrition (Day -1) in all patients treated at Lausanne, CHUV.

OTHER OUTCOMES:
Cancer-specific survival rate | Postoperative time
  Long term overall and cancer-specific survival for bladder cancer patients
Quality of life assessment | 30 and 90 days after surgery
  Assessment of the quality of life after surgery through a questionnaire (EORTC QLQ-C30)
Identification of biomarkers predictive of postoperative complications | Before and after immunonutrition treatement
  Identification of biomarkers predictive of postoperative complications studying the patient's immune and microbiome signature: analysis of immune cells in the blood, analysis of the polyfunctionality of blood T cells, analysis of immune-related proteins in the urine and serum, microbiota analysis, expression of Argininosuccinate synthetase 1

CONTACTS AND LOCATIONS:
Locations (4):
- Switzerland (4):
  - Centre Hospitalier Universitaire Vaudois, CHUV, Lausanne, Canton of Vaud
  - University Hospital of Bern, Bern
  - University Hospital of Geneva, Geneva
  - Hospital of Riviera-Chablais, Rennaz

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Derre L, Crettenand F, Grilo N, Stritt K, Kiss B, Tawadros T, Domingos-Pereira S, Roth B, Cerantola Y, Lucca I. The role of preoperative immunonutrition on morbidity and immune response after cystectomy: protocol of a multicenter randomized controlled trial (INCyst Trial). Trials. 2024 Oct 17;25(1):687. doi: 10.1186/s13063-024-08536-5. PMID 39415282